CLINICAL TRIAL: NCT05037682
Title: Addressing Opioid Use Disorder in the Elderly Through Primary Care Innovation: Pain and Opioid Management in Older Adults
Brief Title: Pain and Opioid Management in Older Adults
Acronym: RISE-OK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12359
Record Dates: First submitted 2021-07-12; First posted 2021-09-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pain, Chronic; Opioid Use Disorder
Keywords: Pain Management; Opioid Use Disorder in Older Adults; Implementation Science; Primary Care Practice Improvement
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: Dissemination and Implementation Research (D&I): Involves assisting primary care practices to address pain and opioid management in older adults. The D&I model also involves Practice Assessment, Academic Detailing, Practice Facilitation, Health Information Technology Support, Performance Feedback and Benchmarking, and a Virtual Learning Community.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Care Practices (Other): Dissemination and Implementation Research
  Interventions: Other: Dissemination and Implementation Research

INTERVENTIONS:
Other: Dissemination and Implementation Research — The study will employ a research and implementation design that attempts to balance scientific rigor, research good practices, primary care implementation preferences and numerous limitations related to the study context. A waitlist-controlled, staggered implementation study will be conducted with three groups of 15 practices introduced to the intervention in 3-month intervals, each baseline overlapping with interim measurements of care quality and process outcomes in concurrent groups in every 3 months, followed by a final data collection at the end of the intervention in months 16 and 17, including baseline measures plus semi-structured interviews. The groups and their sequence will not be randomized, but practice characteristics will be used to distribute them among the three groups based on location, type, size and patient mix to maximize the balance of practices among the groups.

SUMMARY:
The extent and depth of the ongoing opioid crisis are well known and many interventions are under way in the United States and other countries to alleviate its devastating impact on individuals and the society. To address specific challenges of pain and opioid management (POM) in older and vulnerable adults, the investigators will design and implement a multi-faceted, person-centered, and scalable opioid use disorder (OUD) management program in Oklahoma primary care practices. The investigators expect that the rigorously designed and evidence-based program will establish and disseminate innovative solutions for pain and opioid management in high-risk, older and vulnerable populations living with chronic pain. The proposed initiative will help primary care practices optimize pain management approaches in older adults through an integrated and trans-disciplinary application of innovations in multi-modal pain management, pain mechanism-based pharmacotherapy, patient goal-oriented care, implementation science, evidence-based quality improvement methodology, and community-engaged design.

DETAILED DESCRIPTION:
The project's specific aims are:

1. Building upon existing guidelines and tools that the investigators' collaborative has developed and implemented for pain and opioid management (POM), refine and tailor care processes, implementation support strategies, and shared decision support resources to the specific needs of older adults in primary care settings, using a systematic approach, including:

   1. Conduct a rapid, iterative process, through which a diverse healthcare professional expert panel adapts and enhances existing POM approaches and tools to older adult patients (POMOA);
   2. Implement a subsequent formative process, through which a patient and caregiver community advisory board ensures that the tailored POM approach and resources are acceptable, usable, context-sensitive and value-added for older adults and their caregivers; and
   3. Assemble tailored resources to create a POMOA Toolkit from which primary care practices can select sets of resources based on their specific needs, guided by academic detailers and practice facilitators.
2. Over a 2-year period, help a minimum of 36 Oklahoma primary care practices implement a person-centered, goal-oriented, and community-linked approach to pain management, tailored to older adults. The implementation approach will include the following:

   1. Using benchmarking and performance feedback, academic detailing, practice facilitation, and technology support, help practices integrate the tailored POMOA approach and resources into their workflows, focusing on improving patient functioning, self-efficacy, and the optimization of pain management; and
   2. Through ongoing observation and analysis, identify facilitators and barriers to program implementation to accelerate convergence on effective and replicable methods.
3. Conduct a multi-dimensional and comprehensive evaluation of the impact of the RISE-OK program, including the measurement of the following outcomes:

   1. Patient-Centered Outcomes: Patient health-related quality of life and functioning (PROMIS-29), self- efficacy for pain management using a modified Arthritis Self-Efficacy scale (ASES), pain interference (Pain-Enjoyment-General Activity), and functional goal attainment (Goal Attainment Scaling);
   2. Care Quality Outcomes: Patient utilization of opioid medications (morphine milligram equivalents) and alternative therapies in older adults, change in prescribing patterns, and diversification of pharmacological and non-pharmacological pain therapies;
   3. Care Process Outcomes: Impact of the program on practice-level care process outcomes (chronic opioid therapy registry use; systematic chronic opioid therapy visits; pain impact/interference measurement, pain management and risk/benefit conversations; naloxone prescription; tapering practices; patient/caregiver education; shared decision-making; referrals/community service linkages; medication assisted therapy utilization); and
   4. Qualitative Outcomes: Healthcare professional, health system leadership, patient, and caregiver perceptions of the utility, effectiveness and generalizability of the RISE-OK program, explored via semi-structured interviews, exit surveys, and in-depth program implementation process observations.
4. Disseminate innovative approaches and products developed by the RISE-OK project in several ways:

   1. Community-based dissemination (community-based and professional health organizations);
   2. Academic dissemination (presentations, workshops, papers, Agency for Healthcare Research and Quality's communication professionals); Web-based and social networking-based dissemination (e.g., Research-to-Practice Exchange).

ELIGIBILITY:
Inclusion Criteria:

* For the Practice: Deliver primary care services to older adults. Be located in Oklahoma. Be willing to complete a pre- and post-practice characteristic and building blocks of primary care survey. Use an electronic health record.
* For Practice Clinicians: Be an MD, DO, PA, or APRN licensed to practice in Oklahoma. Be willing to complete a pre- and post- practice member survey. Be willing to work with the OPHIC external support personnel to use the performance measures.
* For Practice Staff: Be employed by the practice. Be willing to complete a pre- and post- practice member survey. Be willing to work with the OPHIC external support personnel to use performance measures to optimize pain management approaches in older adults.
* For Practice Patients: Be chronic pain patients aged 60 or older, or may be younger, but vulnerable due to disability, significant functional limitation or social deprivation. Be willing to complete PROMIS-29 surveys, participate in RISE-OK Project activities, and provide feedback on the RISE-OK program.

Exclusion Criteria:

* Practices: Does not provide primary care. Provides only urgent care and does not provide continuity of care or long-term follow-up care. Does not use an electronic health record.
* Clinicians: Do not provide primary care with continuity and chronic care follow-up. Planning to leave practice within the next 12 months, including if the clinician is planning to retire within the next 12 months.
* Practice Staff: Under 18 years of age.
* Patients: Not older adult chronic pain patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life and Functioning: Physical Health Summary Score | Baseline to 17 months
  Change in Patient-Reported Outcomes Measurement Information System Survey (PROMIS-29) Physical Health Summary Score
Health-Related Quality of Life and Functioning: Mental Health Summary Score | Baseline to 17 months
  Change in Patient-Reported Outcomes Measurement Information System Survey (PROMIS-29) Mental Health Summary Score
Morphine Milligram Equivalent (MME) | Baseline to 17 months
  Change in mean opioid Morphine Milligram Equivalent (MMEs) at the practice level

SECONDARY OUTCOMES:
Self-Efficacy | Baseline
  Arthritis Self-Efficacy Scale (ASES) Score. The Arthritis Self-Efficacy Scale has 20 items in 3 subscales: self-efficacy for managing pain (PSE), 5 items; self-efficacy for physical function (FSE), 9 items; and self-efficacy for controlling other systems (OSE), 6 items. Items are rated on a 1 (very uncertain) to 10 (very certain) rating scale. Higher scores indicate greater confidence or self-efficacy.
Self-Efficacy | 17 months
  Arthritis Self-Efficacy Scale (ASES) Score. The Arthritis Self-Efficacy Scale has 20 items in 3 subscales: self-efficacy for managing pain (PSE), 5 items; self-efficacy for physical function (FSE), 9 items; and self-efficacy for controlling other systems (OSE), 6 items. Items are rated on a 1 (very uncertain) to 10 (very certain) rating scale. Higher scores indicate greater confidence or self-efficacy.
Pain-Function Interference | Baseline
  3-item Pain-Enjoyment-General Activity (PEG) score
Pain-Function Interference | Month 5
  3-item Pain-Enjoyment-General Activity (PEG) score
Pain-Function Interference | Month 8
  3-item Pain-Enjoyment-General Activity (PEG) score
Pain-Function Interference | Month 12
  3-item Pain-Enjoyment-General Activity (PEG) score
Pain-Function Interference | Month 17
  3-item Pain-Enjoyment-General Activity (PEG) score
Pain-Related Goal Attainment | Baseline
  Summary of 3-point Pain-Related Goal Attainment Scaling. Patients will rate their Pain-Related Goal Attainment using a 3-category response scale (somewhat less than expected (-1), expected goal achievement (0), and somewhat better than expected (+1).
Pain-Related Goal Attainment | Month 17
  Summary of 3-point Pain-Related Goal Attainment Scaling. Patients will rate their Pain-Related Goal Attainment using a 3-category response scale (somewhat less than expected (-1), expected goal achievement (0), and somewhat better than expected (+1).
Polypharmacy Risk | Baseline
  % of Patients also on psychotropics, sedative-hypnotics, muscle relaxants, or cannabionoids
Polypharmacy Risk | Month 5
  % of Patients also on psychotropics, sedative-hypnotics, muscle relaxants, or cannabionoids
Polypharmacy Risk | Month 8
  % of Patients also on psychotropics, sedative-hypnotics, muscle relaxants, or cannabionoids
Polypharmacy Risk | Month 12
  % of Patients also on psychotropics, sedative-hypnotics, muscle relaxants, or cannabionoids
Polypharmacy Risk | Month 17
  % of Patients also on psychotropics, sedative-hypnotics, muscle relaxants, or cannabionoids
Diversification of Pain Therapy | Baseline
  Number (and Type) of pharmacological and non-pharmacological treatment types
Diversification of Pain Therapy | Month 5
  Number (and Type) of pharmacological and non-pharmacological treatment types
Diversification of Pain Therapy | Month 8
  Number (and Type) of pharmacological and non-pharmacological treatment types
Diversification of Pain Therapy | Month 12
  Number (and Type) of pharmacological and non-pharmacological treatment types
Diversification of Pain Therapy | Month 17
  Number (and Type) of pharmacological and non-pharmacological treatment types
Chronic Opioid Therapy Statistics: Eligible Patients | Baseline
  Number of patients 60+ years of age on chronic opioids
Chronic Opioid Therapy Statistics: Eligible Patients | Month 17
  Number of patients 60+ years of age on chronic opioids
Chronic Opioid Therapy Statistics: Visit Addressing Pain Management | Baseline
  % of patients on chronic opioids that were seen at a visit addressing pain management in the 6 months prior to Baseline.
Chronic Opioid Therapy Statistics: Visit Addressing Pain Management | Month 17
  % of patients on chronic opioids that were seen at a visit addressing pain management in the 6 months prior to Month 17 of the study.
Chronic Opioid Therapy Statistics: Chronic Pain Diagnosis | Baseline
  % of patients on chronic opioids with a chronic pain diagnosis
Chronic Opioid Therapy Statistics: Chronic Pain Diagnosis | Month 17
  % of patients on chronic opioids with a chronic pain diagnosis
Chronic Opioid Therapy Statistics: High Risk Patients | Baseline
  % of patients on chronic opioids with MME>50 and benzo
Chronic Opioid Therapy Statistics: High Risk Patients | Month 17
  % of patients on chronic opioids with MME>50 and benzo

CONTACTS AND LOCATIONS:
Overall Officials: Steven Crawford, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Clinical and Translational Science Institute, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Murthy VH. Ending the Opioid Epidemic - A Call to Action. N Engl J Med. 2016 Dec 22;375(25):2413-2415. doi: 10.1056/NEJMp1612578. Epub 2016 Nov 9. No abstract available. PMID 27959718
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Levy S. Youth and the Opioid Epidemic. Pediatrics. 2019 Feb;143(2):e20182752. doi: 10.1542/peds.2018-2752. Epub 2019 Jan 2. PMID 30602544
- [Background] Huhn AS, Strain EC, Tompkins DA, Dunn KE. A hidden aspect of the U.S. opioid crisis: Rise in first-time treatment admissions for older adults with opioid use disorder. Drug Alcohol Depend. 2018 Dec 1;193:142-147. doi: 10.1016/j.drugalcdep.2018.10.002. Epub 2018 Oct 18. PMID 30384321
- [Background] Jones MR, Novitch MB, Sarrafpour S, Ehrhardt KP, Scott BB, Orhurhu V, Viswanath O, Kaye AD, Gill J, Simopoulos TT. Government Legislation in Response to the Opioid Epidemic. Curr Pain Headache Rep. 2019 May 1;23(6):40. doi: 10.1007/s11916-019-0781-1. PMID 31044343
- [Background] Volkow ND, Collins FS. The Role of Science in Addressing the Opioid Crisis. N Engl J Med. 2017 Jul 27;377(4):391-394. doi: 10.1056/NEJMsr1706626. Epub 2017 May 31. No abstract available. PMID 28564549
- [Background] Volkow ND, Frieden TR, Hyde PS, Cha SS. Medication-assisted therapies--tackling the opioid-overdose epidemic. N Engl J Med. 2014 May 29;370(22):2063-6. doi: 10.1056/NEJMp1402780. Epub 2014 Apr 23. No abstract available. PMID 24758595
- [Background] Liebschutz JM, Xuan Z, Shanahan CW, LaRochelle M, Keosaian J, Beers D, Guara G, O'Connor K, Alford DP, Parker V, Weiss RD, Samet JH, Crosson J, Cushman PA, Lasser KE. Improving Adherence to Long-term Opioid Therapy Guidelines to Reduce Opioid Misuse in Primary Care: A Cluster-Randomized Clinical Trial. JAMA Intern Med. 2017 Sep 1;177(9):1265-1272. doi: 10.1001/jamainternmed.2017.2468. PMID 28715535
- [Background] Parchman ML, Von Korff M, Baldwin LM, Stephens M, Ike B, Cromp D, Hsu C, Wagner EH. Primary Care Clinic Re-Design for Prescription Opioid Management. J Am Board Fam Med. 2017 Jan 2;30(1):44-51. doi: 10.3122/jabfm.2017.01.160183. PMID 28062816
- [Background] West NA, Dart RC. Prescription opioid exposures and adverse outcomes among older adults. Pharmacoepidemiol Drug Saf. 2016 May;25(5):539-44. doi: 10.1002/pds.3934. Epub 2015 Dec 13. PMID 26660909
- [Background] Buckeridge D, Huang A, Hanley J, Kelome A, Reidel K, Verma A, Winslade N, Tamblyn R. Risk of injury associated with opioid use in older adults. J Am Geriatr Soc. 2010 Sep;58(9):1664-70. doi: 10.1111/j.1532-5415.2010.03015.x. PMID 20863326
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Edwards RR, Dworkin RH, Sullivan MD, Turk DC, Wasan AD. The Role of Psychosocial Processes in the Development and Maintenance of Chronic Pain. J Pain. 2016 Sep;17(9 Suppl):T70-92. doi: 10.1016/j.jpain.2016.01.001. PMID 27586832
- [Background] Qadeer RA, Shanahan L, Ferro MA. Chronic disruptive pain in emerging adults with and without chronic health conditions and the moderating role of psychiatric disorders: Evidence from a population-based cross-sectional survey in Canada. Scand J Pain. 2017 Oct;17:30-36. doi: 10.1016/j.sjpain.2017.07.009. Epub 2017 Jul 26. PMID 28850370
- [Background] Nahin RL. Estimates of pain prevalence and severity in adults: United States, 2012. J Pain. 2015 Aug;16(8):769-80. doi: 10.1016/j.jpain.2015.05.002. Epub 2015 May 29. PMID 26028573
- [Background] Hser YI, Mooney LJ, Saxon AJ, Miotto K, Bell DS, Huang D. Chronic pain among patients with opioid use disorder: Results from electronic health records data. J Subst Abuse Treat. 2017 Jun;77:26-30. doi: 10.1016/j.jsat.2017.03.006. Epub 2017 Mar 9. PMID 28476267
- [Background] Saari TI, Ihmsen H, Neuvonen PJ, Olkkola KT, Schwilden H. Oxycodone clearance is markedly reduced with advancing age: a population pharmacokinetic study. Br J Anaesth. 2012 Mar;108(3):491-8. doi: 10.1093/bja/aer395. Epub 2011 Dec 26. PMID 22201184
- [Background] Liukas A, Kuusniemi K, Aantaa R, Virolainen P, Neuvonen M, Neuvonen PJ, Olkkola KT. Plasma concentrations of oral oxycodone are greatly increased in the elderly. Clin Pharmacol Ther. 2008 Oct;84(4):462-7. doi: 10.1038/clpt.2008.64. PMID 19238650
- [Background] Machado-Duque ME, Castano-Montoya JP, Medina-Morales DA, Castro-Rodriguez A, Gonzalez-Montoya A, Machado-Alba JE. Association between the use of benzodiazepines and opioids with the risk of falls and hip fractures in older adults. Int Psychogeriatr. 2018 Jul;30(7):941-946. doi: 10.1017/S1041610217002745. Epub 2017 Dec 10. PMID 29223172
- [Background] Seppala LJ, van de Glind EMM, Daams JG, Ploegmakers KJ, de Vries M, Wermelink AMAT, van der Velde N; EUGMS Task and Finish Group on Fall-Risk-Increasing Drugs. Fall-Risk-Increasing Drugs: A Systematic Review and Meta-analysis: III. Others. J Am Med Dir Assoc. 2018 Apr;19(4):372.e1-372.e8. doi: 10.1016/j.jamda.2017.12.099. Epub 2018 Mar 2. PMID 29402646
- [Background] Gerlach LB, Olfson M, Kales HC, Maust DT. Opioids and Other Central Nervous System-Active Polypharmacy in Older Adults in the United States. J Am Geriatr Soc. 2017 Sep;65(9):2052-2056. doi: 10.1111/jgs.14930. Epub 2017 May 3. PMID 28467623
- [Background] Reid MC, Henderson CR Jr, Papaleontiou M, Amanfo L, Olkhovskaya Y, Moore AA, Parikh SS, Turner BJ. Characteristics of older adults receiving opioids in primary care: treatment duration and outcomes. Pain Med. 2010 Jul;11(7):1063-71. doi: 10.1111/j.1526-4637.2010.00883.x. PMID 20642732
- [Background] Wolff JL, Starfield B, Anderson G. Prevalence, expenditures, and complications of multiple chronic conditions in the elderly. Arch Intern Med. 2002 Nov 11;162(20):2269-76. doi: 10.1001/archinte.162.20.2269. PMID 12418941
- [Background] Wenger NS, Solomon DH, Roth CP, MacLean CH, Saliba D, Kamberg CJ, Rubenstein LZ, Young RT, Sloss EM, Louie R, Adams J, Chang JT, Venus PJ, Schnelle JF, Shekelle PG. The quality of medical care provided to vulnerable community-dwelling older patients. Ann Intern Med. 2003 Nov 4;139(9):740-7. doi: 10.7326/0003-4819-139-9-200311040-00008. PMID 14597458
- [Background] Le Roux C, Tang Y, Drexler K. Alcohol and Opioid Use Disorder in Older Adults: Neglected and Treatable Illnesses. Curr Psychiatry Rep. 2016 Sep;18(9):87. doi: 10.1007/s11920-016-0718-x. PMID 27488204
- [Background] Beaudoin FL, Merchant RC, Clark MA. Prevalence and Detection of Prescription Opioid Misuse and Prescription Opioid Use Disorder Among Emergency Department Patients 50 Years of Age and Older: Performance of the Prescription Drug Use Questionnaire, Patient Version. Am J Geriatr Psychiatry. 2016 Aug;24(8):627-636. doi: 10.1016/j.jagp.2016.03.010. Epub 2016 Apr 1. PMID 27426210
- [Background] Maree RD, Marcum ZA, Saghafi E, Weiner DK, Karp JF. A Systematic Review of Opioid and Benzodiazepine Misuse in Older Adults. Am J Geriatr Psychiatry. 2016 Nov;24(11):949-963. doi: 10.1016/j.jagp.2016.06.003. Epub 2016 Jun 7. PMID 27567185
- [Background] Oh G, Abner EL, Fardo DW, Freeman PR, Moga DC. Patterns and predictors of chronic opioid use in older adults: A retrospective cohort study. PLoS One. 2019 Jan 11;14(1):e0210341. doi: 10.1371/journal.pone.0210341. eCollection 2019. PMID 30633773
- [Background] Kastner M, Hayden L, Wong G, Lai Y, Makarski J, Treister V, Chan J, Lee JH, Ivers NM, Holroyd-Leduc J, Straus SE. Underlying mechanisms of complex interventions addressing the care of older adults with multimorbidity: a realist review. BMJ Open. 2019 Apr 3;9(4):e025009. doi: 10.1136/bmjopen-2018-025009. PMID 30948577
- [Background] Mold J. Goal-Directed Health Care: Redefining Health and Health Care in the Era of Value-Based Care. Cureus. 2017 Feb 21;9(2):e1043. doi: 10.7759/cureus.1043. PMID 28367382
- [Background] Nagykaldi ZJ, Tange H, De Maeseneer J. Moving From Problem-Oriented to Goal-Directed Health Records. Ann Fam Med. 2018 Mar;16(2):155-159. doi: 10.1370/afm.2180. PMID 29531108
- [Background] Purkaple BA, Mold JW, Chen S. Encouraging Patient-Centered Care by Including Quality-of-Life Questions on Pre-Encounter Forms. Ann Fam Med. 2016 May;14(3):221-6. doi: 10.1370/afm.1905. PMID 27184992
- [Background] Reuben DB, Tinetti ME. Goal-oriented patient care--an alternative health outcomes paradigm. N Engl J Med. 2012 Mar 1;366(9):777-9. doi: 10.1056/NEJMp1113631. No abstract available. PMID 22375966
- [Background] Reuben DB, Jennings LA. Putting Goal-Oriented Patient Care Into Practice. J Am Geriatr Soc. 2019 Jul;67(7):1342-1344. doi: 10.1111/jgs.15885. Epub 2019 Mar 18. PMID 30882888
- [Background] Goga JK, Michaels A, Zisselman M, DePaolo A, Khushalani S, Walters JK, Poloway A, Roca R, Kopp M. Reducing opioid use for chronic pain in older adults. Am J Health Syst Pharm. 2019 Apr 8;76(8):554-559. doi: 10.1093/ajhp/zxz025. PMID 31361866
- [Background] Mold JW, Aspy CA, Nagykaldi Z; Oklahoma Physicians Resource/Research Network. Implementation of evidence-based preventive services delivery processes in primary care: an Oklahoma Physicians Resource/Research Network (OKPRN) study. J Am Board Fam Med. 2008 Jul-Aug;21(4):334-44. doi: 10.3122/jabfm.2008.04.080006. PMID 18612060
- [Background] McCormack L, Sheridan S, Lewis M, Boudewyns V, Melvin CL, Kistler C, Lux LJ, Cullen K, Lohr KN. Communication and dissemination strategies to facilitate the use of health-related evidence. Evid Rep Technol Assess (Full Rep). 2013 Nov;(213):1-520. doi: 10.23970/ahrqepcerta213. PMID 24423078
- [Background] Mathis SM, Hagemeier N, Hagaman A, Dreyzehner J, Pack RP. A Dissemination and Implementation Science Approach to the Epidemic of Opioid Use Disorder in the United States. Curr HIV/AIDS Rep. 2018 Oct;15(5):359-370. doi: 10.1007/s11904-018-0409-9. PMID 30069724
- [Background] Dwyer JW, Contreras D, Eschbach CL, Tiret H, Newkirk C, Carter E, Cronk L. Cooperative Extension as a Framework for Health Extension: The Michigan State University Model. Acad Med. 2017 Oct;92(10):1416-1420. doi: 10.1097/ACM.0000000000001640. PMID 28353501
- [Background] Grumbach K, Mold JW. A health care cooperative extension service: transforming primary care and community health. JAMA. 2009 Jun 24;301(24):2589-91. doi: 10.1001/jama.2009.923. No abstract available. PMID 19549977
- [Background] Kaufman A, Boren J, Koukel S, Ronquillo F, Davies C, Nkouaga C. Agriculture and Health Sectors Collaborate in Addressing Population Health. Ann Fam Med. 2017 Sep;15(5):475-480. doi: 10.1370/afm.2087. PMID 28893819
- [Background] Phillips RL Jr, Kaufman A, Mold JW, Grumbach K, Vetter-Smith M, Berry A, Burke BT. The primary care extension program: a catalyst for change. Ann Fam Med. 2013 Mar-Apr;11(2):173-8. doi: 10.1370/afm.1495. PMID 23508605
- [Background] Chou AF, Homco JB, Nagykaldi Z, Mold JW, Daniel Duffy F, Crawford S, Stoner JA. Disseminating, implementing, and evaluating patient-centered outcomes to improve cardiovascular care using a stepped-wedge design: healthy hearts for Oklahoma. BMC Health Serv Res. 2018 Jun 4;18(1):404. doi: 10.1186/s12913-018-3189-4. PMID 29866120
- [Background] Bodenheimer T, Ghorob A, Willard-Grace R, Grumbach K. The 10 building blocks of high-performing primary care. Ann Fam Med. 2014 Mar-Apr;12(2):166-71. doi: 10.1370/afm.1616. PMID 24615313
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Pergolizzi JJV, LeQuang JA. Aging High: Opioid Use Disorder in the Elderly Population. OBM Geriatrics. 2018;3(2):1-. doi: 10.21926/obm.geriatr.1902047.
- [Background] Nagykaldi Z, Mold JW, Robinson A, Niebauer L, Ford A. Practice facilitators and practice-based research networks. J Am Board Fam Med. 2006 Sep-Oct;19(5):506-10. doi: 10.3122/jabfm.19.5.506. PMID 16951300
- [Background] Committee on Integrating Primary Care and Public Health; Board on Population Health and Public Health Practice; Institute of Medicine. Primary Care and Public Health: Exploring Integration to Improve Population Health. Washington (DC): National Academies Press (US); 2012 Mar 28. Available from http://www.ncbi.nlm.nih.gov/books/NBK201594/ PMID 24851288
- [Background] Breslow NE, Clayton DG. Approximate Inference in Generalized Linear Mixed Models. Journal of the American Statistical Association. 1993;88(421). doi: 10.2307/2290687.
- [Background] McCullagh P, Nelder JA. Generalized Linear Models. 2nd ed: Chapman & Hall/CRC Press; 1989.
- [Background] Pinheiro JC, Chao EC. Efficient Laplacian and Adaptive Gaussian Quadrature Algorithms for Multilevel Generalized Linear Mixed Models. Journal of Computational and Graphical Statistics. 2012;15(1):58-81. doi: 10.1198/106186006x96962.
- See also: CDC WONDER Database [Internet] 2017 — https://wonder.cdc.gov/
- See also: Medicare Part D Opioid Prescribing Mapping Tool [Internet] 2017 — https://data.cms.gov/tools